CLINICAL TRIAL: NCT01399554
Title: Exercise as Alcohol Use Disorders Intervention for Non-Treatment Seeking Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: University of Connecticut (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jeremiah Weinstock, Assistant Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R03AA020194 (NIH); 1R03AA020194 (NIH)
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Alcohol-Related Disorders
MeSH Terms: conditions — Alcohol-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Assessment Only (No Intervention)
- Weekly Exercise Counseling Intervention (Experimental)
  Interventions: Behavioral: Motivational Enhancement Therapy plus Contingency Management

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy plus Contingency Management — A combination of two motivational enhancement therapy (MET) sessions focused on increasing exercise spaced two months apart and four months of weekly contingency management (CM) for adhering to specific exercise activities. MET is a client-centered, directive method of enhancing intrinsic motivation to change by exploring and resolving ambivalence, and CM is a behavioral treatment offering individuals tangible reinforcers such as prizes for completion of specific target behaviors.
  Other Names: MET; CM
  Arms: Weekly Exercise Counseling Intervention

SUMMARY:
Alcohol use disorders are common and few individuals with the disorder ever seek help. This study proposes to intervene in a novel way - exercise, as it has many mental and physical health benefits and is an activity that is incompatible with simultaneous alcohol use. If effective, this non-stigmatizing intervention may increase the utility and acceptability of interventions for alcohol use disorders and ultimately increase the number of individuals effectively treated.

DETAILED DESCRIPTION:
About 26 million Americans (8.5%) meet criteria for an alcohol use disorder (AUD; i.e., abuse or dependence), and most with an AUD will not ever seek help. A variety of reasons exist for not seeking help, with stigma and desire to handle the problem on one's own being primary among them. Therefore, offering interventions for AUD that do not stigmatize or require an individual to see a mental health professional may increase the utility and acceptability of AUD interventions and ultimately increase the number of individuals effectively treated. This pilot study evaluates exercise as an AUD intervention. Exercise has been proposed as a potential treatment for AUD due to its numerous mental and physical health benefits. Thirty sedentary non-treatment seeking AUD individuals to be recruited from the community via advertisements. Participants will be given a four month YMCA gym membership and will be randomized to one of two conditions: (1) assessment only (AO), or (2) a combination of two motivational enhancement therapy (MET) sessions focused on increasing exercise spaced two months apart and four months of weekly contingency management (CM) for adhering to specific exercise activities. MET is a client-centered, directive method of enhancing intrinsic motivation to change by exploring and resolving ambivalence, and CM is a behavioral treatment offering individuals tangible reinforcers such as prizes for completion of specific target behaviors. Assessments of all participants will take place at baseline, 2-months (mid-treatment), and 4-months (post-treatment. Results from this pilot study will guide future investigations of exercise as a method for intervening with non-treatment seeking AUD individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-55 years
* English speaking
* Sedentary
* Alcohol-related problems
* Recent heavy drinking episodes
* Blood pressure <165/95 mmHg

Exclusion Criteria:

* Currently receiving or desiring treatment for alcohol problems
* Contraindications for exercise
* Acute psychiatric problems that require immediate treatment
* Obese - class II
* Pregnant or desire to become so in the next several months
* Other substance dependence
* In recovery for pathological gambling

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Monthly drinking frequency | Six months

SECONDARY OUTCOMES:
Monthly Exercise Behavior | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Weinstock J, Petry NM, Pescatello LS, Henderson CE, Nelson CR. Randomized clinical trial of exercise for nontreatment seeking adults with alcohol use disorder. Psychol Addict Behav. 2020 Feb;34(1):65-75. doi: 10.1037/adb0000506. Epub 2019 Aug 19. PMID 31424244